CLINICAL TRIAL: NCT07238192
Title: Augmenting Massed Cognitive Processing Therapy (CPT) to Prevent Suicide Risk Among Patients With PTSD
Acronym: mCPT+CRP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Vermont Medical Center (Other); The University of Texas Health Science Center at San Antonio (Other); C.R.Darnall Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christina Bauder, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HT94252410360; HT94252410360 (Other Grant/Funding Number: U.S. Army Medical Research & Development Command)
Record Dates: First submitted 2025-11-12; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Suicidal Ideation; Suicide Attempt
Keywords: PTSD; Cognitive Processing Therapy; military; suicide; Crisis Response Planning
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Suicidal Ideation; Suicide, Attempted; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Plan (TAU) (Active Comparator): Participants assigned to this arm will receive Safety Planning Treatment as Usual (TAU), a brief, structured intervention commonly used by mental health professionals to help individuals identify warning signs, coping strategies, and sources of support to reduce suicide risk.
  Interventions: Behavioral: Cognitive Processing Therapy
- Crisis Response Plan (CRP) (Experimental): Participants assigned to this arm will receive Crisis Response Planning (CRP), a structured intervention designed to help individuals identify and manage suicidal thoughts and behaviors through a collaborative, personalized plan. CRP uses a procedural format distinct from standard safety planning.
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Regardless of which assignment, participants will receive 10 sessions of Cognitive Processing Therapy (CPT) delivered daily Monday through Friday over two consecutive weeks. In CPT treatment participants will complete symptom checklists and learn a variety of skills to help with symptoms of PTSD.

SUMMARY:
The purpose of this research is to see if Crisis Response Planning (CRP), a brief strategy designed to help people cope effectively with emotional crises, combined with Cognitive Processing Therapy (CPT), a talk treatment for posttraumatic stress disorder (PTSD), will reduce suicidal thoughts and behaviors.

DETAILED DESCRIPTION:
This study is designed to learn whether adding Crisis Response Planning (CRP), a brief, personalized strategy for managing emotional crises, to massed Cognitive Processing Therapy (CPT) can reduce suicidal thoughts and behaviors among military personnel and veterans receiving treatment for posttraumatic stress disorder (PTSD). CPT is a well-established, evidence-based psychotherapy for PTSD, and CRP is an evidence-based intervention shown to reduce suicidal ideation and suicide attempts. By combining these two approaches, this study aims to improve outcomes for individuals who are experiencing both PTSD symptoms and recent suicidal thoughts or behaviors.

We will enroll active-duty service members and veterans who meet criteria for PTSD or subthreshold PTSD and who have experienced active suicidal ideation within the past week or a suicide attempt (actual, aborted, or interrupted) within the past month. Participants will be randomly assigned to one of two treatment conditions:

1. massed CPT plus Crisis Response Planning (CRP)
2. massed CPT plus usual care suicide risk management, which involves a standard safety planning procedure.

All participants will receive 10 daily sessions of massed CPT over two consecutive weeks. The suicide-risk intervention (CRP or usual-care safety planning) is introduced during the intake session and reviewed throughout CPT treatment.

The study has three main goals:

Aim 1 is to determine whether adding CRP to CPT reduces suicide attempts and suicidal ideation more effectively than usual care safety planning. We expect that participants who receive CRP will experience larger and faster reductions in suicidal thoughts and fewer suicide attempts during follow-up.

Aim 2 is to identify early indicators of treatment response and relapse. We will examine whether early improvements in suicide-related symptoms predict changes in suicidal ideation during treatment and whether these markers help identify individuals at higher risk for suicidal behavior after treatment.

Aim 3 is to understand which parts of CRP are most helpful to participants. We will explore how often participants use CRP outside of sessions, which components they find most beneficial, and how these factors relate to reductions in suicidal thinking and behavior.

This study builds on promising preliminary findings. In earlier research conducted by this team, CRP led to faster reductions in suicidal thoughts and fewer suicide attempts than usual care risk-management procedures when paired with massed CPT. Additional analyses have shown that early reductions in suicidal ideation during PTSD treatment may be especially important for long-term recovery from both suicide risk and PTSD symptoms. However, more research is needed to confirm these results in a larger sample and to better understand the mechanisms through which CRP may improve outcomes.

Participants will complete baseline assessments, 10 massed CPT sessions, ecological momentary assessment (EMA) surveys for four weeks, optional booster sessions, and follow-up assessments at 1, 3, 6, 9, and 12 months. The study will take place at the STRONG STAR clinical offices located at the Carl R. Darnall Army Medical Center (CRDAMC) at Fort Hood. Participants may be compensated for completing study assessments, EMA surveys, and other research activities.

By studying both clinical outcomes and early markers of change, this project aims to improve suicide-prevention strategies for military personnel and veterans and provide clinicians with better tools to identify and respond to suicide risk during PTSD treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty service member or veteran aged 18 or older eligible for military medical care.
2. Able to read, write, and speak English.
3. Meeting diagnostic criteria for PTSD or subthreshold PTSD (i.e., meeting diagnostic threshold for 3 of 4 symptom criteria within the past month) on the Clinician Administered PTSD Scale for DSM-5 (CAPS-5).
4. Active suicidal ideation within the past week as assessed by scoring ≥ 1 on Scale for Suicidal Ideation (SSI) item 4 (i.e., active suicidal ideation within the past month) or report an interrupted, aborted, or actual suicide attempt within the preceding month on the Self-Injurious Thoughts and Behaviors Interview-Revised (SITBI-R).
5. Regular use of an iPhone or Android smartphone.

Exclusion Criteria:

1. Inability to comprehend and complete the consent and baseline screening questionnaires.
2. Current suicide or homicide risk meriting crisis intervention.
3. Serious mental health symptoms, such as mania, psychosis, alcohol or substance use disorders warranting immediate clinical attention based on interviewer assessment and clinical judgement.
4. Currently engaged in evidence-based psychotherapy for PTSD (e.g., Cognitive Processing Therapy, Prolonged Exposure Therapy, Written Exposure Therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | From baseline to 12-months follow up
  The PTSD Checklist for the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (PCL-5) is a 20-item self-report measure used to assess PTSD symptom severity and monitor clinical change over time. Each item is rated on a 5-point scale (0 = Not at all to 4 = Extremely), yielding a total score ranging from 0 to 80, with higher scores indicating worse PTSD symptom severity.
Self-Injurious Thoughts and Behaviors Interview-Revised (SITBI-R) | Baseline to 12 months posttreatment
  The Self-Injurious Thoughts and Behaviors Interview-Revised (SITBI-R) is a structured clinical interview assessing the presence and characteristics of suicidal and nonsuicidal thoughts and behaviors. The SITBI-R does not produce a single total score; instead, each item is coded dichotomously as 0 = "No" or 1 = "Yes" to indicate the presence of a given thought or behavior. Higher item values indicate the presence of the self-injurious thought or behavior being assessed.

SECONDARY OUTCOMES:
Scale for Suicide Ideation (SSI) | Baseline through 12 months follow-up
  The Scale for Suicide Ideation is a 21-item self-report measure of past-week or worse-points suicidal ideation. The minimum score is 0, and the maximum score is 42. Higher scores are indicative of more severe suicidal ideation.

CONTACTS AND LOCATIONS:
Overall Officials: Craig J Bryan, Principal Investigator — University of Vermont

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-07-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT07238192/Prot_000.pdf